CLINICAL TRIAL: NCT05730569
Title: Description and Comparison of Biological Vulnerability in Small Vulnerable Newborns Versus Healthy Community Controls in Urban Burkina Faso (DenBalo): Gut Microbiota, Immune System, and Breastmilk Assembly and Development in the First Days and Weeks of Life
Brief Title: Description and Comparison of Biological Vulnerability in Small Vulnerable Newborns Versus Healthy Community Controls in Urban Burkina Faso
Acronym: DenBalo
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Institut de Recherche en Sciences de la Santé (IRSS) (Unknown); Université NAZI BONI (Other); Hasselt University (Other); University of Virginia (Other); University Hospital, Ghent (Other); Cedars-Sinai Medical Center (Other); Sapient Bioanalytics (Unknown); Stanford University (Other); Centre Muraz (Other); University of Manitoba (Other); Manitoba Interdisciplinary Lactation Center (MILC) (Unknown); Agence de Formation, de Recherche & d'Expertise en Santé pour l'Afrique (AFRICSanté) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0500; INV-035474 & INV-036154 (Other Grant/Funding Number: Bill & Melinda Gates Foundation); 050-2022/CEIRES (Other: Comité d'Éthique Institutionnel pour la Recherche en Sciences de la Santé)
Record Dates: First submitted 2023-01-12; First posted 2023-02-16 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Preterm Birth; Low Birth Weight; Small for Gestational Age at Delivery
Keywords: Preterm Birth; Low Birth Weight; Small for Gestational Age; Small Vulnerable Newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Small Vulnerable Newborns: * Low birth weight: <2500g; and/or,
  * Preterm: born between the 34th and 37th week of pregnancy; and/or,
  * Small for Gestational Age: <10 percentile of INTERGROWTH-21st birthweight standards.
- Healthy Community Controls: * Born after the 37th week of pregnancy; and,
  * Birth weight ≥2500g; and,
  * ≥10 percentile of INTERGROWTH-21st birthweight standards.

SUMMARY:
The aim of the DenBalo study is to apply integrated multi-omics methods to examine the biological mechanisms underlying this vulnerability in Small Vulnerable Newborns (SVNs) in LMICs, with the ultimate goal of identifying targeted interventions to reduce morbidity and mortality in this high-risk population. The evidence generated from this project will ultimately help promote healthy pregnancies and the birth of healthy babies.

To achieve this goal, three research objectives are proposed:

1. To describe and compare gut microbiota, immune system and breastmilk components in SVNs versus healthy community controls in urban Burkina Faso.
2. To describe and compare the development of the gut microbiota, the immune system and breastmilk components during the first six months of life in SVNs versus healthy community controls in urban Burkina Faso.
3. To investigate the relationship between the composition of the gut microbiota, the immune system and breastmilk components during the first six months of life in SVNs versus healthy community controls in urban Burkina Faso.

DETAILED DESCRIPTION:
The first days and weeks of life are characterized by a truly impressive cascade of biological processes that drive neonatal growth and development-all of which are crucial to preparing the newborn for life outside the womb.

First, vaginal delivery exposes neonates to an important natural microbial inoculum from the vaginal microbiota in labor and from the maternal intestinal microbiota at birth. Together, these early colonization events lay the foundation for gut microbiota assembly, inform the arrival of subsequent species through microbial interactions, and dictate infant microbiota maturation. A recent study has shown that a handful of bacteria begin colonizing the infant gut within the first days of life, that gut microbes accumulate gradually over time, and that pioneer strains are retained after a month of life. Whether the gut microbial assembly, maturation, and functional potential differs between SVNs versus healthy, community controls, or is coupled to growth and development, remains unresolved.

Secondly, the first days and weeks of life represent a time of heightened vulnerability to infectious disease. Neonatal infections account for a tragic 40% of mortality in children under five years of age. This critical time period is increasingly seen as a key determinant in health over the entire lifespan. A recent study using a high-dimensional, unbiased approach to characterize neonatal immune system development reported a dramatic, purposeful trajectory in the first week of life. While much remains to be explored, what is known is that early microbial colonization is vital to optimal host immune development and protection from disease and that, after birth, the most important determinant of infant gut colonization is breastfeeding. The impacts of preterm birth, low birth weight, or small for gestational age on immune development and function remain enigmatic and the mediating effect of the gut microbiome unknown.

Thirdly, neonatal nutrition plays a vital role in the two aforementioned processes-because breastfeeding both initiates tropic priming of the newborn gut and transfers numerous immunological factors to the baby. However, few studies have explored the synergy between neonatal microbiome and immunome development, and even fewer through the lens of newborn nutrition. Moreover, virtually zero studies include an integrated characterization of these processes in the SVN. Evidence suggests that, compared to mothers of full-term neonates, the colostrum from mothers of preterm newborns has higher protein and fat content, free amino acids, sodium, and bioactive milk components including HMOs, cytokines, and lactoferrin. But because few studies have evaluated the association between early milk composition and infant growth and development, it is unclear which components are most imperative for a healthy gut microbiota and a robust immune system, particularly in the SVN.

Major advances in systems biology approaches allowing for unbiased, integrated analyses of high-dimensional -omic databases have provided the critical bioinformatic toolkit required to address these questions. Indeed, the ground has never been more fertile for a step-change in commitment to high-impact research on neonatal microbiome and immunome development and the synergy with newborn nutrition.

ELIGIBILITY:
INCLUSION CRITERIA

* Fundal height between 24 and 27 cm
* Woman living in the health zone of Accart-Ville, Colma 1 or Farakan
* Woman not planning to give birth or move outside the study area in the first 6 months of the infant's life
* Gestational age between 24 weeks 0 completed day and 29 weeks 6 days (ultrasound)
* Monofetal pregnancy without visible malformation
* Woman agreeing to give her informed consent to participate in the study
* Delivery of a live birth
* Vaginal birth
* Absence of severe infectious pathology, severe pneumopathy or respiratory distress in the neonate
* Neonates who did not receive corticosteroids or antibiotics at birth

For Small Vulnerable Newborns (SVNs):

* Low birth weight: <2500g; and/or,
* Preterm: born between the 34th and 37th week of pregnancy; and/or,
* Small for Gestational Age: <10 percentile of INTERGROWTH-21st birthweight standards.

For healthy community controls:

* Neonate born after the 37th week of pregnancy; and,
* Birth weight >2500g; and,
* ≥10 percentile of INTERGROWTH-21st birthweight standards; and,
* Possible match with a SVN neonate already recruited into the study.

EXCLUSION CRITERIA

* Fundal height <24 cm or >27 cm
* Woman living outside the sanitary zone of the Accart-Ville, Colma 1 or Farakan
* Woman planning to give birth outside the study area or to move from it within the first 6 months of the infants's life
* Gestational age <24 weeks or ≥30 weeks (ultrasound)
* Multi-fetal pregnancy
* Malformation visible on ultrasound
* Cesarean delivery
* Neonate with severe infectious disease, severe pneumopathy or respiratory distress
* Neonate who received corticosteroids or antibiotics just after birth

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of all pregnant women at the beginning of the third trimester of their pregnancy attending regular antenatal consultations (ANC) at Accart-Ville, Colma 1 or Farakan health centers.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Differential abundances of bacterial genera in the infant gut microbiota | to be assessed at on days 3, 7, 14, 30, 60, 180 of life
  Shotgun metagenomic sequencing

SECONDARY OUTCOMES:
Infant gut microbiota α and β diversity | to be assessed at on days 3, 7, 14, 30, 60, 180 of life
  Shotgun metagenomic sequencing
Infant plasma immunophenotyping | to be assessed at birth and on days 1, 3, 5, 7, 30, 60 of life
  Flow cytometry
Infant plasma chemokine and cytokine analyses | to be assessed at birth and on days 1, 3, 5, 7, 30, 60 of life
  Electrochemiluminescence and the MSD V-PLEX Human Biomarker 54-Plex Kit
Maternal breastmilk component* profiling | on days 3, 7, 14, 30, 60 of life
  *Components include macronutrients, micronutrients, oligosaccharides, growth factors, immunoglobulins, cytokines, metabolites, microbes, and proteins.

OTHER OUTCOMES:
Differential abundance of bacterial populations of pregnant or lactating woman (PLW) fecal microbiota | to be assessed within 28-30 weeks of gestation, within 33-34 weeks of gestation, on days 7, 14, 30, 60 and 180 of life
  Shotgun metagenomic sequencing
PLW Infant fecal microbiota α and β diversity | to be assessed within 28-30 weeks of gestation, within 33-34 weeks of gestation, on days 7, 14, 30, 60 and 180 of life
  Shotgun metagenomic sequencing
PLW fecal enteropathogens | to be assessed within 28-30 weeks of gestation, within 33-34 weeks of gestation, on days 30 and 180 of life
  TaqMan Array Card (TAC) qPCR to detect 62 infection targets of interest, including viruses, bacteria, protozoa and helminths.
Infant fecal enteropathogens | to be assessed within 28-30 weeks of gestation, within 33-34 weeks of gestation, on days 30 and 180 of life
  TaqMan Array Card (TAC) qPCR to detect 62 infection targets of interest, including viruses, bacteria, protozoa and helminths.
Maternal plasma immunophenotyping | to be assessed at birth
  Flow cytometry
Maternal plasma chemokine and cytokine analyses | to be assessed at birth
  Electrochemiluminescence and the MSD V-PLEX Human Biomarker 54-Plex Kit
Black carbon exposure in umbilical cord arterial blood | to be assessed at birth
  White-light generation under femtosecond pulsed illumination
Placental DNA adductiomics | to be assessed at birth
  Hybrid Quadrupole Orbitrap MS (Q-Exactive™) high-resolution mass spectrometry (HRMS)
Relative telomere length (TL) in umbilical cord arterial blood | to be assessed at birth
  qPCR
Infant untargeted metabolomics on capillary whole blood | to be assessed at birth, on days 1, 3, 5, 7, 14, 30 and 60 of life
  Modified Agilent RapidFire 360 sample injector coupled to a high-resolution Agilent 6545B liquid chromatography Quadrupole Time-of-Flight (LC/Q-TOF) next-generation rapid liquid chromatography-mass spectrometry (rLC-MS)
Infant untargeted plasma proteomics | to be assessed at birth, on days 1, 3, 5, 7, 14, 30 and 60 of life
  Harmonized Orbitrap Exploris™ liquid chromatography-mass spectrometry (LC-MS)
Infant multiple mycotoxin profiling on capillary whole blood | to be assessed at birth, on days 7, and 14 of life
  Liquid Chromatography Tandem Mass Spectrometry (LC-MS/MS)
Maternal untargeted capillary whole blood metabolomics | to be assessed at birth
  Modified Agilent RapidFire 360 sample injector coupled to a high-resolution Agilent 6545B liquid chromatography Quadrupole Time-of-Flight (LC/Q-TOF) next-generation rapid liquid chromatography-mass spectrometry (rLC-MS)
Maternal untargeted plasma proteomics | to be assessed at birth
  Harmonized Orbitrap Exploris™ liquid chromatography-mass spectrometry (LC-MS)
Maternal multiple mycotoxin profiling on capillary whole blood | to be assessed at birth
  Liquid Chromatography Tandem Mass Spectrometry (LC-MS/MS)
PLW shotgun vaginal metagenomics | to be assessed 29-30 weeks of gestation, 33-34 weeks of gestation and at birth
  Shotgun metagenomic sequencing
Breastmilk volume intake | to be assessed on days 1, 3, 4, 13 and 14 of life
  "Dose-to-mother" deuterium oxide dilution
Differential abundances of bacterial genera in the infant gut microbiota | to be assessed at birth and on days 1, 2, 4, 5, 6 of life
  Shotgun metagenomic sequencing
Infant gut microbiota α and β diversity | to be assessed at birth and on days 1, 2, 4, 5, 6 of life
  Shotgun metagenomic sequencing
Maternal breastmilk component* profiling | to be assessed at birth and on days 1, 3, 5 of life
  Shotgun metagenomic sequencing
Vaginal cytokines | to be assessed at 29-30 weeks of gestation
  Multi-plex assay

CONTACTS AND LOCATIONS:
Overall Officials: Trenton Dailey-Chwalibóg, MPH, PhD, Principal Investigator — University Ghent; Carl Lachat, MEng, PhD, Principal Investigator — University Ghent
Locations (1):
- Agence de Formation, de Recherche et d'Expertise en Santé pour l'Afrique (AFRICSanté), Bobo-Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
All the data collected during the DenBalo study will be pseudonymised (i.e., identifable data can still be linked to patient files by means of a code) and the key to the codes will only be accessible to the principal investigators, or his/her representative.
  The collected pseudonymised data as well as the collected biological samples can be shared with other (future) researchers for future research projects and studies, exclusively in the context of the same disease/pathology or similar (i.e., in the interest of research on maternal, newborn and child health). This will be done within a strictly legal framework and in compliance with international laws on the protection of personal data.
  Only anonymized data will be used in any type of documentation, reports or publications (in the medical scientific literature and/or at medical conferences).
  Personal patient data will be stored for at least 25 years after the end of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be on embargo for a period of 18 months post study implementation.
Access Criteria: Upon reasonable request.

REFERENCES:
- [Background] Bennike TB, Fatou B, Angelidou A, Diray-Arce J, Falsafi R, Ford R, Gill EE, van Haren SD, Idoko OT, Lee AH, Ben-Othman R, Pomat WS, Shannon CP, Smolen KK, Tebbutt SJ, Ozonoff A, Richmond PC, van den Biggelaar AHJ, Hancock REW, Kampmann B, Kollmann TR, Levy O, Steen H. Preparing for Life: Plasma Proteome Changes and Immune System Development During the First Week of Human Life. Front Immunol. 2020 Oct 20;11:578505. doi: 10.3389/fimmu.2020.578505. eCollection 2020. PMID 33329546
- [Background] Bhutta ZA, Black RE. Global maternal, newborn, and child health--so near and yet so far. N Engl J Med. 2013 Dec 5;369(23):2226-35. doi: 10.1056/NEJMra1111853. No abstract available. PMID 24304052
- [Background] Bittinger K, Zhao C, Li Y, Ford E, Friedman ES, Ni J, Kulkarni CV, Cai J, Tian Y, Liu Q, Patterson AD, Sarkar D, Chan SHJ, Maranas C, Saha-Shah A, Lund P, Garcia BA, Mattei LM, Gerber JS, Elovitz MA, Kelly A, DeRusso P, Kim D, Hofstaedter CE, Goulian M, Li H, Bushman FD, Zemel BS, Wu GD. Bacterial colonization reprograms the neonatal gut metabolome. Nat Microbiol. 2020 Jun;5(6):838-847. doi: 10.1038/s41564-020-0694-0. Epub 2020 Apr 13. PMID 32284564
- [Background] Bode L. Human milk oligosaccharides: every baby needs a sugar mama. Glycobiology. 2012 Sep;22(9):1147-62. doi: 10.1093/glycob/cws074. Epub 2012 Apr 18. PMID 22513036
- [Background] Chu H, Mazmanian SK. Innate immune recognition of the microbiota promotes host-microbial symbiosis. Nat Immunol. 2013 Jul;14(7):668-75. doi: 10.1038/ni.2635. PMID 23778794
- [Background] Funkhouser LJ, Bordenstein SR. Mom knows best: the universality of maternal microbial transmission. PLoS Biol. 2013;11(8):e1001631. doi: 10.1371/journal.pbio.1001631. Epub 2013 Aug 20. PMID 23976878
- [Background] Granger CL, Embleton ND, Palmer JM, Lamb CA, Berrington JE, Stewart CJ. Maternal breastmilk, infant gut microbiome and the impact on preterm infant health. Acta Paediatr. 2021 Feb;110(2):450-457. doi: 10.1111/apa.15534. Epub 2020 Sep 16. PMID 33245565
- [Background] Jost T, Lacroix C, Braegger CP, Rochat F, Chassard C. Vertical mother-neonate transfer of maternal gut bacteria via breastfeeding. Environ Microbiol. 2014 Sep;16(9):2891-904. doi: 10.1111/1462-2920.12238. Epub 2013 Sep 3. PMID 24033881
- [Background] Kollmann TR, Kampmann B, Mazmanian SK, Marchant A, Levy O. Protecting the Newborn and Young Infant from Infectious Diseases: Lessons from Immune Ontogeny. Immunity. 2017 Mar 21;46(3):350-363. doi: 10.1016/j.immuni.2017.03.009. PMID 28329702
- [Background] Lee AH, Shannon CP, Amenyogbe N, Bennike TB, Diray-Arce J, Idoko OT, Gill EE, Ben-Othman R, Pomat WS, van Haren SD, Cao KL, Cox M, Darboe A, Falsafi R, Ferrari D, Harbeson DJ, He D, Bing C, Hinshaw SJ, Ndure J, Njie-Jobe J, Pettengill MA, Richmond PC, Ford R, Saleu G, Masiria G, Matlam JP, Kirarock W, Roberts E, Malek M, Sanchez-Schmitz G, Singh A, Angelidou A, Smolen KK; EPIC Consortium; Brinkman RR, Ozonoff A, Hancock REW, van den Biggelaar AHJ, Steen H, Tebbutt SJ, Kampmann B, Levy O, Kollmann TR. Dynamic molecular changes during the first week of human life follow a robust developmental trajectory. Nat Commun. 2019 Mar 12;10(1):1092. doi: 10.1038/s41467-019-08794-x. PMID 30862783
- [Background] Ma J, Li Z, Zhang W, Zhang C, Zhang Y, Mei H, Zhuo N, Wang H, Wang L, Wu D. Comparison of gut microbiota in exclusively breast-fed and formula-fed babies: a study of 91 term infants. Sci Rep. 2020 Sep 25;10(1):15792. doi: 10.1038/s41598-020-72635-x. PMID 32978424
- [Background] Makino H, Kushiro A, Ishikawa E, Kubota H, Gawad A, Sakai T, Oishi K, Martin R, Ben-Amor K, Knol J, Tanaka R. Mother-to-infant transmission of intestinal bifidobacterial strains has an impact on the early development of vaginally delivered infant's microbiota. PLoS One. 2013 Nov 14;8(11):e78331. doi: 10.1371/journal.pone.0078331. eCollection 2013. PMID 24244304
- [Background] Makino H, Kushiro A, Ishikawa E, Muylaert D, Kubota H, Sakai T, Oishi K, Martin R, Ben Amor K, Oozeer R, Knol J, Tanaka R. Transmission of intestinal Bifidobacterium longum subsp. longum strains from mother to infant, determined by multilocus sequencing typing and amplified fragment length polymorphism. Appl Environ Microbiol. 2011 Oct;77(19):6788-93. doi: 10.1128/AEM.05346-11. Epub 2011 Aug 5. PMID 21821739
- [Background] Melville JM, Moss TJ. The immune consequences of preterm birth. Front Neurosci. 2013 May 21;7:79. doi: 10.3389/fnins.2013.00079. eCollection 2013. PMID 23734091
- [Background] Mueller NT, Shin H, Pizoni A, Werlang IC, Matte U, Goldani MZ, Goldani HAS, Dominguez-Bello MG. Delivery Mode and the Transition of Pioneering Gut-Microbiota Structure, Composition and Predicted Metabolic Function. Genes (Basel). 2017 Dec 4;8(12):364. doi: 10.3390/genes8120364. PMID 29207565
- [Background] Nayak S, Welling J, Burd I. Maternal Immunomodulation Therapy for Prevention of Preterm Birth and Prematurity-Related Morbidity: The New Era of Immuno-Perinatology. Curr Pharm Des. 2017;23(40):6125-6131. doi: 10.2174/1381612823666170926102615. PMID 28950816
- [Background] Underwood MA. Human milk for the premature infant. Pediatr Clin North Am. 2013 Feb;60(1):189-207. doi: 10.1016/j.pcl.2012.09.008. Epub 2012 Oct 18. PMID 23178065